CLINICAL TRIAL: NCT05741073
Title: Outcome Research of a European Registry Platform on Real-world Treatment Data of Patients with Advanced NMSC
Status: Recruiting | Type: Observational
Sponsor: EuMelaReg gGmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: Euro-NMSC
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Basal Cell Carcinoma; Cutaneous Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- resected HR-cSCC: Patients with resected HR-cSCC (Cohort 1) receiving only postoperative radiotherapy or watchful waiting
- advanced cSCC: Patients with advanced cSCC who are not candidates for curative surgery/radiation in routine clinical practice (Cohort 2)
- advanced BCC: Patients with advanced BCC who are not candidates for curative surgery/radiation in routine clinical practice (Cohort 3)

SUMMARY:
This current registry study will analyze real-world data to address questions about disease characteristics and treatment patterns in NMSC patients based on the European NMSC-Registry. The overall objective is to describe characteristics, management and treatment outcomes for patients presenting with advanced NMSC (cSCC/BCC) or HR-cSCC in routine clinical practice, independent of treatments used across different European regions.

DETAILED DESCRIPTION:
Skin cancer is one of the most common cancers worldwide, and the most frequent cancer in the white population. Incidence rates of NMSC are increasing, partly attributable to more outdoor leisure activities and aging population. Among NMSC, basal cell carcinoma (BCC) and cutaneous squamous cell carcinoma (cSCC) are the most predominant histologic subtypes. Real-world data especially those systematically recorded in registries are limited. With limited resources, many cancer databases do not register all primary NMSCs. For advanced patients with NMSC, the EUMelaReg consortium (EMR) introduces a registry specific for NMSC across Europe (EMR-NMSC) which brings together national registries and operates as a higher-level registry. The aim of this registry is to collect real-world data of the available diagnosis and treatment pattern of advanced NMSC patients at a European level. Data of the EMR NMSC-Registry can be used for specific pre-defined analyses regarding drugs, availability and affordability of various treatments for different patient populations, data on health-related resource utilization, outcome data, and risk factors.

Quality management Study participating sites are responsible for recording and verifying the accuracy of subject data.

A data management plan (DMP) will be in place which describes the life cycle of the study data from the collection to archiving, including all measures to ensure that the data remain available, usable and comprehensible. It includes rules and regulations for e.g. data validation, data processing, medical coding, quality review procedures and archiving of study documentation. National and international data protection laws as well as regulations on registries will be followed.

Data validation Detailed information on checks for completeness, accuracy, plausibility and validity are given in the data validation plan (DVP). The computerized handling of the data by the service provider may generate requests to which the participating site needs to respond by confirming or modifying the data questioned.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years at index date
2. Patients documented in the European NMSC-registry fulfilling EMR quality standard
3. Patients with resected HR-cSCC (Cohort 1) receiving only postoperative radiotherapy or watchful waiting OR Patients with advanced cSCC who are not candidates for curative surgery/radiation in routine clinical practice (Cohort 2) OR Patients with advanced BCC who are not candidates for curative surgery/radiation in routine clinical practice (Cohort 3)

Exclusion Criteria:

1. Patients receiving treatment within a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with documentation of advanced diagnosis of cSCC/ BCC or with HR-cSCC since AUG 2019 and who fulfill the inclusion and exclusion criteria described below will be included in this registry. Enrollment into all 3 cohorts will be performed concurrently. All patients will be treated according to specifications stated in the respective local/European guidelines of the drugs administered in clinical routine.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Real-world demographics in routine clinical practice | min. 2 years up to max 5 years of observation
  To capture real-world demographics in routine clinical practice, independent of treatment used across different European regions in patients with advanced cSCC, advanced BCC, and completely resected HR-cSCC.

SECONDARY OUTCOMES:
Tumor characteristics | min. 2 years up to max 5 years of observation
  To describe tumor characteristics (pathology, site and stage)
Treatment patterns | min. 2 years up to max 5 years of observation
  To evaluate treatment patterns in patients with advanced cSCC, advanced BCC, and completely resected HR-cSCC in routine practice
Overall survival | min. 2 years up to max 5 years of observation
  To characterize overall survival (OS) from initiation of treatment in the advanced stage (for HR-cSCC: from date of surgery) to date of death due to any cause
Adverse drug reactions | min. 2 years up to max 5 years of observation
  To described adverse drug reactions (ADRs)
Treatment discontinuation | min. 2 years up to max 5 years of observation
  Reason for treatment discontinuation
Time to progression (TTP) - for advanced BCC only | min. 2 years up to max 5 years of observation
  Time to progression (TTP) of first and second line treatment for advanced BCC defined as time from start of treatment to date of progression based on physician's assessment or death due to aBCC.
Time to progression (TTP) - for advanced cSCC | min. 2 years up to max 5 years of observation
  Time to progression (TTP) for advanced cSCC defined as time from start of treatment to date of progression based on physician's assessment or death due to cSCC.
Time to next treatment (TTNT) - for advanced cSCC, advanced BCC only | min. 2 years up to max 5 years of observation
  Time to next treatment (TTNT) defined as the time from the date of treatment initiation in the advanced stage until the next line of treatment.
Time to treatment discontinuation (TTD) - for advanced cSCC, advanced BCC only | min. 2 years up to max 5 years of observation
  Time to treatment discontinuation (TTD), defined as the interval between start of treatment and its permanent discontinuation or death.
Progression free survival (PFS) - for advanced cSCC, advanced BCC only | min. 2 years up to max 5 years of observation
  Progression free survival (PFS) from start of treatment in the advanced stage to progression based on physician's assessment or death due to any cause.
Overall response rate (ORR) - for advanced cSCC, advanced BCC only | min. 2 years up to max 5 years of observation
  Overall response rate (ORR) during first line/second line treatment defined as the proportion of patients with CR or PR as best response according to physician's routine method.
Time to recurrence (TTR) | min. 2 years up to max 5 years of observation
  For resected high-risk cSCC, defined as AJCC 8th edition T class of T3 tumor or any resected N-positive regional disease only:
  Time to recurrence (TTR) defined as time from date of R0-surgery to date of recurrence or tumour related death.
Disease Free Survival (DFS) | min. 2 years up to max 5 years of observation
  For resected high-risk cSCC, defined as AJCC 8th edition T class of T3 tumor or any resected N-positive regional disease only:
  Disease Free Survival (DFS) defined as period from complete resection to date of relapse or death of any cause.
Freedom from distant recurrence (FFDR) | min. 2 years up to max 5 years of observation
  For resected high-risk cSCC, defined as AJCC 8th edition T class of T3 tumor or any resected N-positive regional disease only:
  Freedom from distant recurrence (FFDR) defined as time from date of R0-surgery to date of occurrence of a distant metastasis.
Freedom from locoregional recurrence (FFLRR) | min. 2 years up to max 5 years of observation
  For resected high-risk cSCC, defined as AJCC 8th edition T class of T3 tumor or any resected N-positive regional disease only:
  Freedom from locoregional recurrence (FFLRR) defined as time from date of R0-surgery to date of occurrence of a local relapse or locoregional metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ (Universitair Ziekenhuis) Brüssel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No